CLINICAL TRIAL: NCT07376070
Title: The Role of Inflammatory Biomarkers in Preventing Deep Sternal Wound Infections After Sternotomy
Status: Active, not recruiting | Type: Observational
Sponsor: Levan Nebieridze (Other)
Responsible Party: Sponsor-Investigator, Levan Nebieridze, Junior physician, cardiac surgery, Tbilisi State Medical University
Organization: Tbilisi State Medical University (Other)
Other Study IDs: TbilisiSMU
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Deep Sternal Infection; Diabete Mellitus; Mediastinitis
MeSH Terms: conditions — Diabetes Mellitus; Mediastinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this observational study is to reveal blood biomarkers that will have prognostic significance in terms of the development of deep wound infection following sternotomy. As for the practical significance of the study, blood biomarkers correlated with deep wound infections can be used to prevent the development of wound infections in the postoperative period. Based on this, it is possible to formulate an algorithm for preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* deep sternal wound infection

Exclusion Criteria:

* bilateral internal thoracic artery graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from Georgia, who undergo cardiac surgery operation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
change in pre and postoperative inflammatory biomarker levels associated with development of deep sternal wound infection within 1 month | within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Tbilisi State Medical University, Tbilisi
  - Bokhua memorial cardiovascular center, Tbilisi